CLINICAL TRIAL: NCT01752582
Title: BuMA OCT Study(A Comparative Evaluation of BuMA Stent and of EXCEL Stent in Terms of the Extent of Neointima Formation at 3 Months After Implantation Using OCT)
Brief Title: BuMA OCT Study(A Comparative Evaluation of the Extent of Neointima Formation at 3 Months After Implantation Using OCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: version1.1
Record Dates: First submitted 2012-12-07; First posted 2012-12-19 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Heart Disease; Stable Angina Pectoris; Unstable Angina Pectoris; Silent Myocardial Ischemia
Keywords: BuMA; EXCEL; OCT; stent; neointima formation
MeSH Terms: conditions — Coronary Disease; Angina, Stable; Angina, Unstable; Neointima

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BuMA stent (Other): This study will enroll a total of 70 patients in Fuwai Hospital.All patients will be randomly assigned two groups(in a 1:1 ratio).
  BuMA stent Arm:About 35 patients will undergoing implantation of BuMA stent.All of the patients will receive 6 months dual antiplatelet therapy and they will be followed (at the outpatient clinic) for up to 2 years. The follow-up visits will be conducted at 3 months(including angiographic/OCT investigation), 6 months, 1 and 2 years post PCI,in order to observe the Primary Endpoint and Secondary Endpoints.
  Interventions: Device: BuMA stent
- EXCEL stent (Other): This study will enroll a total of 70 patients in Fuwai Hospital.All patients will be randomly assigned two groups(in a 1:1 ratio).
  EXCEL stent Arm:About 35 patients will undergoing implantation of EXCEL stent.All of the patients will receive 6 months dual antiplatelet therapy and they will be followed (at the outpatient clinic) for up to 2 years. The follow-up visits will be conducted at 3 months(including angiographic/OCT investigation), 6 months, 1 and 2 years post PCI,in order to observe the Primary Endpoint and Secondary Endpoints.
  Interventions: Device: EXCEL stent

INTERVENTIONS:
Device: BuMA stent — About 35 patients will undergoing implantation of BuMA stent and receive 6 months dual antiplatelet therapy.
  Arms: BuMA stent
Device: EXCEL stent — About 35 patients will undergoing implantation of EXCEL stent and receive 6 months dual antiplatelet therapy.
  Arms: EXCEL stent

SUMMARY:
The objective of this study is a comparative evaluation of BuMA stent and of EXCEL stent in terms of the extent of neointima formation at 3 months after implantation using OCT.

This is a prospective, single center, randomized, open-label, non-inferiority study, which will enroll a total of 70 patients in Fuwai Hospital.All patients will be randomly assigned undergoing implantation of BuMA stent or EXCEL stent (in a 1:1 ratio). If non-inferiority was met, superiority test will be planned.

DETAILED DESCRIPTION:
About 70 patients with clinical evidence of ischemic heart disease and / or a positive functional study and documented stable angina pectoris (Canadian cardiovascular society classification (CCS)1, 2, 3 or 4), or documented silent ischemia in de-novo, native, previously unstented vessel in Fuwai Hospital,will be randomly assigned undergoing implantation of BuMA stent or EXCEL stent (in a 1:1 ratio).

All of the patients will receive 6 months dual antiplatelet therapy and they will be followed (at the outpatient clinic) for up to 2 years. The follow-up visits will be conducted at 3 months (including angiographic/OCT investigation), 6 months, 1 and 2 years post percutaneous coronary intervention(PCI),in order to observe the Primary Endpoint and Secondary Endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years.
* Evidence of myocardial ischemia without raised troponin (e.g. stable or unstable angina, silent ischemia demonstrated by positive territorial functional study).
* The patient has a planned intervention of up to four de novo lesions, in different epicardial vessels.
* Lesion(s) must have a visually estimated diameter stenosis of ≥50% and <100%.
* Reference Vessel Diameter(RVD) must be between 2.5-4.0 mm
* Written informed consent.
* The patient and the patient's physician agree to the follow-up visits including angiographic follow-up and OCT controls at 3 months.

Exclusion Criteria:

* Evidence of ongoing acute myocardial infarction in ECG prior to procedure.
* Left ventricular ejection fraction(LVEF) <30%.
* Documented or suspected liver disease (including laboratory evidence of hepatitis).
* Known renal insufficiency (e.g. estimated glomerular filtration rate(eGFR) <60 ml/kg/m2 or serum creatinine level of >2.5 mg/dL, or subject on dialysis).
* History of bleeding diathesis or coagulopathy.
* The patient is a recipient of a heart transplant.
* Known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel and ticlopidine), sirolimus or stainless steel.
* Other medical illness (e.g. cancer, neurological deficiency) or known history of substance abuse (alcohol etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy.
* Pregnant or breastfeeding woman or woman in fertile period not taking adequate contraceptives

OCT exclusion criteria

* Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in suboptimal imaging or excessive risk of complication from placement of an OCT catheter
* Total occlusion or thrombolysis in myocardial infarction(TIMI) flow 0, prior to wire crossing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the percentage of the struts'neointimal coverage (%) at 3 months follow-up by OCT assessment. | three months after surgery
  The primary outcome measure is the percentage of the struts'neointimal coverage (%) at 3 months follow-up by OCT assessment.

SECONDARY OUTCOMES:
Neointimal hyperplasia area/volume | three months after surgery
  It will be measure the neointimal hyperplasia area/volume at 3 months follow-up by OCT assessment.
Mean/Minimal Stent diameter/area/volume | three months after surgery
  It will be measure the Mean/Minimal stent diameter/area/volume at 3 months follow-up by OCT assessment.
Mean/Minimal Lumen diameter/area/volume | three months after surgery
  It will be measure the Mean/Minimal Lumen diameter/area/volume at 3 months follow-up by OCT assessment.
Mean/maximal thickness of the struts coverage | three months after surgery
  It will be measure the Mean/maximal thickness of the struts coverage at 3 months follow-up by OCT assessment.
Incomplete strut apposition | three months after surgery
  It will be measure the incomplete strut apposition at 3 months follow-up by OCT assessment.
Minimal Lumen Diameter(MLD) and Diameter stenosis percentage(%DS) post procedure and at 3 months | three months after surgery
Late Lumen Loss at 3 months | three months after surgery
Binary Restenosis (DS ≥50%) at 3 months | three months after surgery
  All measurements will be made of the in-stent, in-segment, proximal and distal stent margins.
Acute success rate | up to 7 days after surgery
  It includes the device success,lesion success and procedural success.
Device-oriented Composite Endpoints and its individual components at 3 months | three months after surgery
  Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, Myocardial Infarction(MI) not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Device-oriented Composite Endpoints and its individual components at 6 months | six months after surgery
  Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Device-oriented Composite Endpoints and its individual components at 1 year | one year after surgery
  Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Device-oriented Composite Endpoints and its individual components at 2 years | 2 years after surgery
  Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Stent thrombosis according to the ARC definitions at 3 months | three months after surgery
Stent thrombosis according to the ARC definitions at 6 months | six months after surgery
Stent thrombosis according to the ARC definitions at 1 year | one year after surgery
Stent thrombosis according to the ARC definitions at 2 years | 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yang Y Jin, president, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Science
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China